CLINICAL TRIAL: NCT02632097
Title: Randomized Prospective Double-Blinded Study of Histoacryl™Mesh Fixation Compared to Conventional Non-absorbable Suture Fixation During Lichtenstein Hernioplasty
Brief Title: Histoacryl™ vs. Suture for Mesh Fixation in Lichtenstein Hernioplasty: A Randomized Prospective Double-Blinded Study
Acronym: Histoacryl1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Plató (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Histoacryl1
Record Dates: First submitted 2015-12-13; First posted 2015-12-16 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; mesh fixation; glue; cyanoacrylate; Lichtenstein; ambulatory surgery
MeSH Terms: conditions — Hernia, Inguinal | interventions — Enbucrilate; Sutures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Histoacryl (Experimental): Intervention: Lichtenstein Hernioplasty with Histoacryl™(cyanoacrylate glue 0.5 ml) for mesh fixation (Optilene™ mesh 60 g/m2 (B. Braun))
  Interventions: Procedure: Lichtenstein Hernioplasty with Histoacryl
- Suture (Experimental): Intervention: Lichtenstein Hernioplasty with Sutures (polypropylene 2/0) to fix the Optilene™ mesh 60 g/m2 (B. Braun)
  Interventions: Procedure: Lichtenstein Hernioplasty with Sutures

INTERVENTIONS:
Procedure: Lichtenstein Hernioplasty with Histoacryl — Procedure/Surgery: Lichtenstein Hernioplasty with Histoacryl:
  0.5 ml of cyanoacrylate glue is used for mesh fixation
  Arms: Histoacryl
Procedure: Lichtenstein Hernioplasty with Sutures — Procedure/Surgery: Lichtenstein Hernioplasty with Sutures: non-absorbable suture (polypropylene 2/0) is used for mesh fixation Other Name: prolene 2-0
  Arms: Suture

SUMMARY:
This is a prospective, randomized double-blinded study to find out if mesh fixation with n-butyl-2-cyanoacrylate (NBCA) are more painless than conventional mesh fixation with sutures in inguinal hernia operation (Lichtenstein procedure) in day-case surgery. Our hypothesis is that glue fixation is safe, simple and fast method compared to conventional Lichtenstein technique.

DETAILED DESCRIPTION:
Hypothesis:

1. To use glue (instead of sutures) for mesh fixation during open hernioplasty causes a lower immediate postoperative pain.
2. The use of Histoacryl is associated to a lower postoperative complications rate.
3. The use of Histoacryl is not associated to a higher hernia recurrence rate.

Methods:

350 patients with inguinal hernia undergone Lichtenstein operation in day-case surgery setting. Mesh fixation is performed using 2 methods: cyanoacrylate glue: Histoacryl™ (n=175: Group H), and non-absorbable sutures: polypropylene 2/0 (n=175: Group S). Operative time and pain scores, immediate postoperative outcome are followed 1, 7, 30 days and 1 and 5 years postoperatively.

Surgeon doesn't know previously which fixation method will be used in each patient. This method (glue or sutures) is decided intraoperatively, when mesh is placed, using a blind randomization code (www.randomizer.org) Patients are discharged (day-case surgery) if adequate pain control, oral tolerance and spontaneous diuresis is achieved, and after examination by the surgeon in order to discard immediate complications. Postoperative oral treatment is prescribed to patients of both groups: dexketoprofen 25 mg/8 h + paracetamol 1 gr/8.

Follow-up is performed at the medical office by a blind observer (third surgeon) who didn't participate in the surgical procedure, at 1 day, 7 days, 30 days, 1 year and annually thereafter. Pain is measured using a VAS scale (0-10).

Operative data (including operating time, complications, hospital stay, etc.), early and late complications, acute and chronic pain and recurrence rate will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* unilateral inguinal hernia
* primary hernia

Exclusion Criteria:

* femoral hernia
* recurrent inguinal hernia
* immunosuppression (including corticosteroids, radiotherapy, chemotherapy)
* chronic renal failure (hemodialysis)
* active infection
* pregnancy
* allergy to polypropylene
* patient's refusal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Acute Postoperative Pain | 30 days
  pain scores (VAS 0-10) after surgery
Operating Time | 30 days
  operating time needed to perform hernioplasty

SECONDARY OUTCOMES:
Postoperative Complications | 30 days
  Complications related to procedure and assessed according to Clavien-Dindo Classification
Early Recurrence Rate | 1 year
  Inguinal hernia recurrence rate after 1 year follow-up
Chronic Pain | 1 year
  Pain scores (0-10) after 1-year follow-up
Late Recurrence Rate | 5 years
  Inguinal hernia recurrence rate after 5 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Hoyuela, MD, Principal Investigator — Hospital Plató
Locations (1):
- Hospital Plató, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lichtenstein IL, Shulman AG, Amid PK, Montllor MM. The tension-free hernioplasty. Am J Surg. 1989 Feb;157(2):188-93. doi: 10.1016/0002-9610(89)90526-6. PMID 2916733
- [Background] Amid PK, Lichtenstein IL. Long-term results and current status of the Lichtenstein open tension-free hernioplasty. Hernia 1998; 2: 89-94
- [Result] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Derived] Hoyuela C, Juvany M, Carvajal F, Veres A, Troyano D, Trias M, Martrat A, Ardid J, Obiols J, Lopez-Cano M. Randomized clinical trial of mesh fixation with glue or sutures for Lichtenstein hernia repair. Br J Surg. 2017 May;104(6):688-694. doi: 10.1002/bjs.10488. Epub 2017 Feb 20. PMID 28218406